CLINICAL TRIAL: NCT04551352
Title: An Open-Label, Multicenter, Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7293583, A TYRP1-Targeting CD3 T-Cell Engager, in Participants With Metastatic Melanoma
Brief Title: A Study of RO7293583 in Participants With Unresectable Metastatic Tyrosinase Related Protein 1 (TYRP1)-Positive Melanomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP42169; 2020-000793-18 (EudraCT Number)
Record Dates: First submitted 2020-08-26; First posted 2020-09-16 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Cutaneous Melanoma; Uveal Melanoma; Mucosal Melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — tocilizumab; obinutuzumab; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I: Single Participant Cohorts (IV) (Experimental): Part I is a dose escalation in single participant cohorts. RO7293583 will be administered intravenously (IV) every three weeks (Q3W). The starting dose will be 0.045mg and the maximum dose explored will be 1.5mg.
  Interventions: Drug: RO7293583; Drug: Tocilizumab
- Part II: Multiple Participant Cohorts (IV/SC) (Experimental): Multiple ascending dose-escalation of RO7293583 in multiple participant cohorts: The starting-dose for the initiation of the IV dose-escalation will be determined by Part I and RO7293583 will be administered IV or SC every 3 weeks. Dose-escalation will be undertaken based on safety until determination of the MTD or the highest safe dose if MTD is not reached. Fractionated, step up or subcutaneous dosing may be implemented. The maximum dose explored will be 600mg IV and 160mg SC.
  Interventions: Drug: RO7293583; Drug: Tocilizumab; Drug: Obinutuzumab; Drug: Adalimumab

INTERVENTIONS:
Drug: RO7293583 — RO7293583 will be administered at a dose and per schedule as specified for the respective cohort.
Drug: Tocilizumab — Tocilizumab will be administered as required for the management of severe cytokine release syndrome (CRS).
  Other Names: Actemra
Drug: Obinutuzumab — If implemented, it will be given either on D-7 or D-7 and D-6.
  Other Names: Gazyva
  Arms: Part II: Multiple Participant Cohorts (IV/SC)
Drug: Adalimumab — If implemented, it will be given as a single dose approximately 6 days prior to the first dose of RO7293583.
  Other Names: Humira
  Arms: Part II: Multiple Participant Cohorts (IV/SC)

SUMMARY:
This is a first-in-human, multi-center clinical study to determine the safety, Maximum Tolerated Dose (MTD) and/or Optimal Biological Dose (OBD) as well as the optimal schedule for intravenous (IV) and/or subcutaneous (SC) administrations of RO7293583 with or without obinutuzumab pretreatment, in participants with unresectable metastatic TYRP1-positive melanomas who have progressed on standard of care (SOC) treatment, are intolerant to SOC, or are non-amenable to SOC. This study will include an initial single participant dose-escalation part one followed by a multiple participant dose-escalation part two with the possibility of expansion.

ELIGIBILITY:
Inclusion Criteria:

* Participants with unresectable stage III or stage IV cutaneous melanoma or participants with unresectable, metastatic uveal or mucosal melanoma for whom SOC is not available or who are intolerant or non-amenable to SOC.
* Participants with cutaneous melanoma need to have known BRAF status.
* Radiologically measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Availability of a representative tumor specimen that is suitable for determination of TYRP1 status by means of central testing.
* For participants in Part II, willingness to provide mandatory on-treatment biopsies.
* Life expectancy (in the opinion of the Investigator) of ≥12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Absence of rapid disease progression, threat to vital organs or non-irradiated lesions > 2 cm in diameter at critical sites.
* All acute toxic effects of any prior radiotherapy, chemotherapy, targeted or checkpoint inhibitor therapy, or surgical procedure must have resolved to Grade ≤1 or returned to baseline, except for alopecia (any grade), for Grade 2 clinically controlled sequelae of immune-related toxicities related to checkpoint inhibitor therapy like adrenal insufficiency and hypopituitarism, and for Grade 2 peripheral neuropathy.
* Adequate hematological, liver and renal function.

Exclusion Criteria:

* Participants with a history or clinical evidence of central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days before screening.
* Participants with another invasive malignancy in the last 2 years.
* Active, acute, or chronic inflammatory diseases of the skin affecting more than 5% of the body surface area. History of Stevens-Johnson syndrome, toxic epidermal necrolysis, or drug rash with eosinophilia and systemic symptoms.
* Participants with defects in the Bruch's membrane of the eye or at risk of such defects. Participants with a history of recurrent uveitis or medical conditions that are associated with frequent uveitis.
* History of or existing damage to inner ear.
* Uncontrolled hypertension.
* Significant cardiovascular disease.
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial, parasitic or other infection, or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks prior to the start of drug administration.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug.
* Major surgery or significant traumatic injury <28 days prior to the first RO7293583 administration or anticipation of the need for major surgery during study treatment.
* Last dose of checkpoint inhibitors, targeted therapies, chemotherapy, immunostimulating or immunosuppressive therapy or other investigational drug <28 days prior to the first RO7293583 administration.
* Prior treatment with a T-cell engaging drug

Specific Exclusion Criteria if Pre-treatment with Obinutuzumab is Implemented:

* Known human immunodeficiency virus (HIV)
* History of progressive multifocal leukoencephalopathy.
* Active Tuberculosis (TB) requiring treatment within 3 years prior to baseline.
* Latent TB diagnosed during Screening.
* Positive test results for human T-lymphotropic virus 1.

Specific Exclusion Criteria if Pre-treatment with Adalimumab is Implemented:

* History of untreated tuberculosis or untreated active infection with mycobacterium tuberculosis.
* Known hypersensitivity to any of the components of adalimumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | From Day 1 of Cycle 1 up to Day 1 of Cycle 3 (each cycle is 21 days)
  Dose-Limiting Toxicities (DLTs) were reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0), except for Cytokine release syndrome (CRS), which will be graded based on the American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Percentage of Participants with Adverse Events (AEs) | Baseline up to 60 days after last RO7293583 treatment (up to 14 months)
  An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of RO7293583 | Up to 14 months
Time of Maximum Concentration (Tmax) of RO7293583 | Up to 14 months
Minimum Concentration (Cmin) of RO7293583 | Up to 14 months
SC Bioavailability (F) of RO7293583 | Up to 14 months
Clearance (CL) or Apparent Clearance (CL/F) of RO7293583 | Up to 14 months
Volume of Distribution at Steady State (Vss) of RO7293583 | Up to 14 months
Area Under the Curve (AUC) of RO7293583 | Up to 14 months
Percentage of Participants with Anti-Drug Antibodies (ADAs) to RO7293583 | From baseline until 60 days after last RO7293583 dose (up to 14 months).
Change from Baseline in RO7293583 ADA Titer | From baseline until 60 days after last RO7293583 dose (up to 14 months).
Objective Response Rate (ORR) | Baseline up to 13 months
  ORR is defined as the percentage of participants with confirmed objective response (OR). Confirmed OR is defined as complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Disease Control Rate (DCR) | Baseline up to 13 months
  DCR is defined as the percentage of participants with CR, PR, or stable disease (SD). Per RECIST v1.1, CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum on study. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline, or the appearance of one or more new lesions.
Duration of Response (DOR) | Baseline up to 13 months
  DOR is defined as the time from the first occurrence of documented OR to disease progression, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Progression-Free Survival (PFS) | Baseline up to 24 months.
  PFS is defined as the time from Cycle 1, Day 1 to the first occurrence of disease progression, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Overall Survival (OS) | Baseline up to 24 months.
  OS is defined as the time from Cycle 1, Day 1 to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Thomas Jefferson University Hospital;Medical Oncology, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Peter Maccallum Cancer Institute; Clinical Trial Unit, Melbourne, Victoria, Australia
- Belgium (2):
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
- Canada (2):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- Herlev Hospital; Afdeling for Kræftbehandling, Herlev, Denmark
- Spain (4):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Vall d´Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Clinica Universidad de Navarra Madrid; Servicio de Oncología, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spreafico A, Couselo EM, Irmisch A, Bessa J, Au-Yeung G, Bechter O, Svane IM, Sanmamed MF, Gambardella V, McKean M, Callahan M, Dummer R, Klein C, Umana P, Justies N, Heil F, Fahrni L, Opolka-Hoffmann E, Waldhauer I, Bleul C, Staack RF, Karanikas V, Fowler S. Phase 1, first-in-human study of TYRP1-TCB (RO7293583), a novel TYRP1-targeting CD3 T-cell engager, in metastatic melanoma: active drug monitoring to assess the impact of immune response on drug exposure. Front Oncol. 2024 Mar 21;14:1346502. doi: 10.3389/fonc.2024.1346502. eCollection 2024. PMID 38577337